CLINICAL TRIAL: NCT05212831
Title: Portable Oxygen Concentrator (POC) Versus Standard of Care in Patients With Long-COVID Cognitive Impairment: a Randomized Crossover Exploratory Pilot Study.
Brief Title: Portable Oxygen Concentrator (POC) Versus Standard of Care in Long-COVID: Randomized Crossover Exploratory Pilot Study.
Acronym: RESTORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inogen Inc. (Industry)
Collaborators: The Montreal Health Innovations Coordinating Center (MHICC) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: INO-01
Record Dates: First submitted 2022-01-21; First posted 2022-01-28 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard of Care (SOC) (No Intervention): SOC is defined as the patient symptoms or complications based treatment.
- Portable Oxygen Concentrator (Experimental): Inogen One® G4 Portable Oxygen Concentrator (POC) is used on a prescriptive basis by subjects requiring supplemental oxygen. It supplies a high concentration of oxygen and is used with a nasal cannula which channels oxygen from the concentrator to the subject.
  Inogen One® G4 is designed to provide a flow of high purity oxygen. Inogen One® G4 may be used in home, institution, vehicle and various mobile environments.
  Interventions: Device: Inogen One® G4

INTERVENTIONS:
Device: Inogen One® G4 — Inogen One® G4 will be used for a minimum of 3h per day at Setting 3 during the intervention period.
  Arms: Portable Oxygen Concentrator

SUMMARY:
A prospective, open label, randomized, crossover, pilot, exploratory study to describe the effect of the Inogen One® G4 POC on brain hypoxia, peripheral oxygen saturation and cognitive function in adults with longterm- COVID.

DETAILED DESCRIPTION:
After a 2-week screening/baseline evaluation, participants will be randomized in a 1:1 allocation ratio to one of the following 2 sequences: 1) portable oxygen concentrator (POC) for a first 2-week period followed by standard of care (SOC) for a second 2-week period or 2) SOC for a first 2-week period followed by POC for a second 2-week period. There will be a washout period of one week between the two treatment periods. A total of 10 subjects will be enrolled per sequence.

ELIGIBILITY:
Inclusion Criteria:

1. Ability and willingness to give written informed consent prior to any study-specific screening procedures and to comply with the requirements of the study
2. Male or female, aged ≥ 18 years of age
3. Diagnosed with Long-COVID
4. Patient self-reported concerns regarding cognitive functioning or recent diagnosis of COVID-19 related cognitive impairment
5. MoCA test scores ranging from 13 to 25/30 at screening
6. Oxygen saturation SpO2 ≤ 93 % on fingertip pulse oximetry and/or < 60% on brain NIRS, at rest or during effort and/ or 10% relative decrease in brain saturation during exercise as compared to baseline value at screening
7. Ability to perform exercise treadmill test at screening
8. Tolerability of pulsed oxygen (O2) therapy delivered by POC at screening
9. Willingness and ability to wear POC.

Exclusion Criteria:

1. Contraindication to the use of POC including allergy to cannula material
2. Pregnancy or planning to become pregnant during the study
3. Non-COVID-related cause for cognitive impairment (such as Parkinson's disease, multiple sclerosis, Alzheimer's disease, stroke, brain tumor, or dementia)
4. Subjects with respiratory infection at screening or randomization and/or acute bronchitis requiring antibiotics at the time of randomization or expected during the treatment
5. Participation in other interventional clinical trial within 30 days of randomization or expect to participate in any other investigational clinical trial during the conduct of this trial
6. Subjects who should be excluded in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
COVID-19 related brain hypoxia and peripheral oxygen saturation | 14+/-3 days
  To describe the effect of the Inogen One® G4 POC on COVID-19 related brain hypoxia and peripheral oxygen saturation
VO2max during cardiopulmonary exercise test | 14+/-3 days
  To describe the effect of the Inogen One® G4 POC on VO2max during cardiopulmonary exercise test
MoCA test | 14+/-3 days
  To describe the effect of the Inogen One® G4 POC on Cognitive performance using the MoCA test
Other neuropsychological tests | 14+/-3 days
  To describe the effect of the Inogen One® G4 POC on Cognitive health assessments using other neuropsychological tests

SECONDARY OUTCOMES:
Functional status | 14+/-3 days
  To describe the effect of the Inogen One® G4 POC on post-COVID functional status
Anxiety, mood, and subjective cognitive impairment | 14+/-3 days
  To describe the effect of the Inogen One® G4 POC on anxiety, mood, and subjective cognitive impairment
Pulmonary function | 14+/-3 days
  To describe the effect of the Inogen One® G4 POC on the post COVID-19 pulmonary function
Safety outcomes | 14+/-3 days
  To determine the safety outcomes of the Inogen One® G4 POC in this subject population

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Montreal Heart Institute, Montreal, Quebec
  - Centre ÉPIC de l'Institut de cardiologie de Montréal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No